CLINICAL TRIAL: NCT06791746
Title: Compound Staphylococcal Lysostaphin Versus Chlorhexidine Mouthrinse for the Prophylaxis of Oral Mucositis in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation: a Randomized, Controlled, Non-inferiority Clinical Tria
Brief Title: Compound Staphylococcal Lysostaphin Vs. Chlorhexidine Mouthrinse for Oral Mucositis in Patients Undergoing Allo-HSCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, XY Zhou, Head Nurse, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019.1114
Record Dates: First submitted 2025-01-13; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Stem Cell Transplant Complications; Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- compound Staphylococcal lysostaphin mouthrinse (Experimental): Patients in the compound Staphylococcal lysostaphin mouthrinse group received OM prophylaxis by sequential gargling with 15 ml of sodium bicarbonate mouthrinse and 15 ml of compound Staphylococcal lysostaphin mouthrinse.
  Interventions: Drug: compound Staphylococcal lysostaphin mouthrinse
- chlorhexidine mouthrinse (Active Comparator): The chlorhexidine mouthrinse group followed the same protocol using 15 ml of sodium bicarbonate mouthrinse and 15 ml of chlorhexidine mouthrinse.
  Interventions: Drug: chlorhexidine mouthrinse

INTERVENTIONS:
Drug: compound Staphylococcal lysostaphin mouthrinse — Lysostaphin is a proteolytic enzyme produced by a specific species of Staphylococcus, uniquely capable of cleaving the cross-linking pentaglycine bridges within the cell walls of Staphylococcus aureus.
  Arms: compound Staphylococcal lysostaphin mouthrinse
Drug: chlorhexidine mouthrinse — Chlorhexidine mouthrinse offers a cost-effective prophylactic approach to preventing OM.
  Arms: chlorhexidine mouthrinse

SUMMARY:
Oral mucositis (OM) is a common complication in patients receiving myeloablative conditioning allogeneic hematopoietic stem cell transplantation (allo-HSCT). Chlorhexidine mouthrinse offers a cost-effective prophylactic approach to preventing OM, yet its use is hampered by issues like tooth discoloration, unpleasant taste, and pain on ulcerated surfaces, leading to reduced patient compliance. This study aims to demonstrate the non-inferior efficacy of a compound Staphylococcal lysostaphin mouthrinse to that of chlorhexidine mouthrinse in reducing OM occurrence in patients receiving myeloablative conditioning allo-HSCT.

DETAILED DESCRIPTION:
This study aims to demonstrate the non-inferior efficacy of a compound Staphylococcal lysostaphin mouthrinse (Xinjingjie Mouthrinse®) to that of chlorhexidine mouthrinse in reducing OM occurrence in patients receiving myeloablative conditioning allo-HSCT. It also seeks to observe patient treatment adherence and pain, so as to provide evidence for the appropriate OM prevention and management measures in clinical practice. This randomized, controlled, non-inferiority clinical trial was conducted at the Bone Marrow Transplant Center, the First Affiliated Hospital of Medical College, Zhejiang University from January 2020 to December 2021.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant hematological diseases who are undergoing allogeneic hematopoietic stem cell transplantation (HSCT) from fully matched sibling donors, unrelated donors, or haploidentical related donors.
* The conditioning regimen is myeloablative, specifically the BUCY regimen (comprising cytarabine, busulfan, and cyclophosphamide), with methotrexate used for graft-versus-host disease (GVHD) prophylaxis. The dosage of cytarabine is ≥4.0g/m²/day, busulfan is ≥3.2mg/m²/day, and cyclophosphamide is ≥1.8g/m²/day.
* There are no restrictions on age or gender.
* Patients voluntarily agree to participate in this trial.

Exclusion Criteria:

* Patients with an expected survival time of less than one month;
* Patients who have already developed oral mucositis (OM) prior to conditioning;
* Patients undergoing autologous stem cell transplantation;
* Patients receiving a non-myeloablative conditioning regimen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
cumulative incidence of oral mucositis | Time from day 0 to the day of neutrophil engraftment (usually within 30 days after transplantation).

SECONDARY OUTCOMES:
severity of oral mucositis | Time from day 0 to the day of neutrophil engraftment (usually within 30 days after transplantation).
  The severity of OM was assessed according to the WHO grading criteria.
the onset time of oral mucositis | Time from day 0 to the day of neutrophil engraftment (usually within 30 days after transplantation).
oral pain | Time from day 0 to the day of neutrophil engraftment (usually within 30 days after transplantation).
  Oral pain was evaluated using the Numeric Rating Scale (NRS), ranging from 0 to 10, with higher numbers indicating greater pain intensity.
compliance with mouth rinsing | Time from day 0 to the day of neutrophil engraftment (usually within 30 days after transplantation).
  Compliance was measured by the average daily frequency of mouthrinse use.
the number of days new analgesics are used due to OM | Time from day 0 to the day of neutrophil engraftment (usually within 30 days after transplantation).
time to neutrophil engraftment | Time from day 0 to the day of neutrophil engraftment (usually within 30 days after transplantation).
  Neutrophil engraftment was defined as three consecutive days with a neutrophil count >0.5×10e9/L.

CONTACTS AND LOCATIONS:
Locations (1):
- Bone marrow transplantation center, the First Affiliated Hospital of Medical College, Zhejiang University, Hangzhou, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No